CLINICAL TRIAL: NCT07362212
Title: Validity, Reliability, and Clinical Correlates of Virtual Reality Adaptations of the 4-meter Walk Test, Five Times Sit-to-stand Test, and Timed up and go Test in Older Adults
Brief Title: Virtual Reality-Based Functional Mobility Tests in Older Adults
Status: Not yet recruiting | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Mehmet Kaan ALTUNOK, Lecturer, Selcuk University
Other Study IDs: SelcukU_PT_OP_VR_ADAPTATION_1
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Functional Mobility; Virtual Reality-Based Functional Assessment
Keywords: Older Adults; Functional Mobility; Virtual Reality; 4-Meter Walk Test; Five-Times Sit-to-Stand Test; Timed Up and Go Test; Validity and Reliability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older Adults: Older adults undergoing conventional and virtual reality-based assessments of functional mobility, balance, and lower extremity function, including the 4-Meter Walk Test, Five-Times Sit-to-Stand Test, and Timed Up and Go Test, to evaluate validity, reliability, and clinical correlates.
  Interventions: Other: Clinical Assessments

INTERVENTIONS:
Other: Clinical Assessments — Participants will perform virtual reality-based adaptations of the 4-Meter Walk Test, Five-Times Sit-to-Stand Test, and Timed Up and Go Test using an immersive virtual reality application developed for the Meta Quest 3 platform. The virtual environment digitally replicates the conventional test setups and protocols, and performance outcomes are automatically recorded by the system. Virtual reality-based assessments will be compared with conventional clinical tests and repeated to evaluate validity, reliability, and clinical correlates.

SUMMARY:
Objective assessment of mobility, balance, and lower extremity function in older adults is of great importance in both clinical practice and scientific research. For this purpose, performance-based tests that can be administered in a short time, are easily repeatable, and have high clinical practicality are widely preferred. These tests provide valuable information about older adults' ability to perform activities of daily living, levels of functional independence, and risk of falls, thereby contributing significantly to both diagnostic processes and treatment planning.

One of these tests, the 4-Meter Walk Test (4MWT), is among the simplest and most reliable methods used to assess walking speed in older adults. Gait speed is considered a strong indicator of functional capacity and overall health status in older individuals and is also used as a critical parameter for predicting mortality, morbidity, hospitalization rates, and duration of independent living. Therefore, due to its short administration time, high repeatability, and clinical validity, the 4MWT has become one of the standard assessment tools in the field of geriatrics.

Another frequently used assessment tool, the Five-Times Sit-to-Stand Test (5xSTS), is based on measuring the time required for an individual to consecutively stand up from and sit down on a chair five times. This test is closely associated with lower extremity muscle strength, functional independence, and the ability to maintain activities of daily living. In addition, the 5xSTS test is an important clinical tool for identifying muscle weakness and mobility limitations in older adults with a history of falls. Owing to its short administration time, lack of requirement for specialized equipment, and ease of understanding, it is widely used in both clinical settings and field studies.

In addition, the Timed Up and Go (TUG) test is considered one of the gold standard methods for the assessment of functional mobility. The test is simple to administer: the time required for an individual to stand up from a chair, walk a specified distance, turn around, and return to sit down is measured. The TUG test not only assesses mobility but is also a reliable and valid method for predicting balance impairments and fall risk. Given that falls represent a major health concern in older adults, data obtained from the TUG test provide valuable guidance for both clinicians and researchers.

In recent years, virtual reality (VR)-based assessment methods have attracted increasing attention due to their potential to provide a safe, motivating, and standardized environment, particularly for older adults. In this study, the Meta Quest 3 virtual reality headset and controllers will be used to implement VR-based functional tests. The Meta Quest 3 device features a resolution of 2064 × 2208 pixels per eye, a maximum refresh rate of 120 Hz, and a six-degrees-of-freedom (6 DoF) inside-out tracking system. The device tracks participants' head and body movements in real time and accurately reflects them within the virtual environment. This system does not require external sensors and automatically provides positional tracking in the virtual space. Previous studies have demonstrated that VR applications can produce valid and reliable outcomes when used as digital adaptations of functional tests. However, the validity and reliability of VR adaptations of the 4MWT, 5xSTS, and TUG tests in older adults have not yet been systematically investigated.

The rationale of this study is to determine whether VR-based short performance tests can serve as a safer, more easily repeatable, and potentially more accessible alternative to conventional clinical assessments. The findings of this study are expected to provide important evidence supporting the use of VR technology in clinical practice for the assessment of mobility and balance in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older,
* Ability to ambulate independently (assistive devices permitted),
* Cognitive ability sufficient to communicate and follow instructions,
* Provision of written informed consent.

Exclusion Criteria:

* Acute cardiopulmonary disease,
* Uncontrolled hypertension,
* History of lower extremity surgery or fracture within the past 6 months,
* Severe cognitive impairment preventing cooperation with testing procedures,
* Determination by a healthcare professional that participation is unsafe for safety-related reasons.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community-dwelling adults aged 65 years and older who are able to ambulate independently (with or without assistive devices) and can communicate and follow test instructions.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
4-Meter Walk Test - Virtual Reality (4MWT-VR) | Baseline and 5-7 days
  This outcome measure will be used to assess gait speed using a virtual reality-based adaptation of the 4-Meter Walk Test. Walking speed will be automatically calculated by the system. Validity will be evaluated by comparison with the conventional 4-Meter Walk Test, and reliability will be assessed using repeated measurements performed 5-7 days apart.
Five-Times Sit-to-Stand Test - Virtual Reality (5xSTS-VR) | Baseline and 5-7 days
  This outcome measure will be used to assess lower extremity functional performance using a virtual reality-based adaptation of the Five-Times Sit-to-Stand Test. Test duration will be automatically recorded. Validity and reliability will be evaluated by comparison with the conventional test and repeated measurements.
Timed Up and Go Test - Virtual Reality (TUG-VR) | Baseline and 5-7 days
  This outcome measure will be used to assess functional mobility using a virtual reality-based adaptation of the Timed Up and Go test. Test completion time will be automatically recorded by the system. Validity and reliability will be examined through comparison with the conventional Timed Up and Go test and repeated measurements.

SECONDARY OUTCOMES:
4-Meter Walk Test - Conventional | Baseline
  The conventional 4-Meter Walk Test will be administered to assess gait speed and will be used as a reference measure for concurrent validity analyses.
Five-Times Sit-to-Stand Test - Conventional | Baseline
  The conventional Five-Times Sit-to-Stand Test will be used to assess lower extremity muscle strength and functional mobility and will serve as a reference for validity analyses.
Timed Up and Go Test - Conventional | Baseline
  The conventional Timed Up and Go test will be administered to assess functional mobility and fall risk and will be used as a reference for concurrent validity analyses.
Lower Extremity Muscle Strength | Baseline
  Lower extremity muscle strength will be measured using standardized clinical methods and will be examined for its relationship with virtual reality-based performance test outcomes.
Physical Activity Level (International Physical Activity Questionnaire - Short Form, IPAQ-SF) | Baseline
  Physical activity level will be assessed using the International Physical Activity Questionnaire - Short Form (IPAQ-SF) and will be analyzed as a clinical correlate of virtual reality-based functional performance tests.

CONTACTS AND LOCATIONS:
Overall Officials: İsmail ÖZSOY, Assoc. Prof. Dr., Study Chair — Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Türkiye; Gülşah ÖZSOY, Assist. Prof. Dr., Study Chair — Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Türkiye; Zehra KORKUT, Assist. Prof. Dr., Study Chair — Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Türkiye; Mehmet A GÜLER, PhD, Study Chair — Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Türkiye; Yasemin GEDİKLİ ERTÜRK, MSc. in PT, Study Chair — Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Türkiye; Muhammed İ KODAK, Assist. Prof. Dr., Study Chair — Kırşehir Ahi Evran University, School of Physical Therapy and Rehabilitation, Kırşehir, Türkiye; Ahmet ÇİZMECİOĞLU, Assoc. Prof. Dr., Study Chair — Selcuk University, Faculty of Medicine, Department of Internal Medicine, Konya, Türkiye
Locations (1):
- Selcuk University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saglam M, Arikan H, Savci S, Inal-Ince D, Bosnak-Guclu M, Karabulut E, Tokgozoglu L. International physical activity questionnaire: reliability and validity of the Turkish version. Percept Mot Skills. 2010 Aug;111(1):278-84. doi: 10.2466/06.08.PMS.111.4.278-284. PMID 21058606
- [Background] Maden C, Gozacan Karabulut D, Bagci B. Validity and reliability of an immersive virtual reality adaptation of the 6-minute pegboard and ring test. Hand Surg Rehabil. 2025 Feb;44(1):101981. doi: 10.1016/j.hansur.2024.101981. Epub 2024 Oct 30. PMID 39486588
- [Background] Barry E, Galvin R, Keogh C, Horgan F, Fahey T. Is the Timed Up and Go test a useful predictor of risk of falls in community dwelling older adults: a systematic review and meta-analysis. BMC Geriatr. 2014 Feb 1;14:14. doi: 10.1186/1471-2318-14-14. PMID 24484314
- [Background] Bohannon RW. Sit-to-stand test for measuring performance of lower extremity muscles. Percept Mot Skills. 1995 Feb;80(1):163-6. doi: 10.2466/pms.1995.80.1.163. PMID 7624188
- [Background] Studenski S, Perera S, Patel K, Rosano C, Faulkner K, Inzitari M, Brach J, Chandler J, Cawthon P, Connor EB, Nevitt M, Visser M, Kritchevsky S, Badinelli S, Harris T, Newman AB, Cauley J, Ferrucci L, Guralnik J. Gait speed and survival in older adults. JAMA. 2011 Jan 5;305(1):50-8. doi: 10.1001/jama.2010.1923. PMID 21205966